CLINICAL TRIAL: NCT07208539
Title: A Prospective, Double-cohort, Multicenter, Phase II Study of Gemcitabine and Albumin Paclitaxel in Combination With PD-L1 Antibodies Followed by Liposomal Irinotecan Combined With Oxaliplatin, 5-FU/LV and PD-L1 Antibodies as Conversion Therapy for Borderline Resectable/Local Advanced Pancreatic Cancer
Brief Title: AG Followed by FOLFIRINOX Both Combined With PD-L1 Antibodies as a Conversion Therapy for Borderline Resectable and Locally Advanced Pancreatic Cancer.
Acronym: ZSPAC-14
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZSPAC-14
Record Dates: First submitted 2025-09-28; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — folfirinox

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sequential therapy (Experimental)
  Interventions: Drug: Treatment: AG & anti-PD-L1 + FOLFIRINOX & anti-PD-L1

INTERVENTIONS:
Drug: Treatment: AG & anti-PD-L1 + FOLFIRINOX & anti-PD-L1 — The cohort A (borderline resectable) and cohort B (locally advanced) both received treatment with gemcitabine, albumin paclitaxel (administered on days 1, 8, and 15, with 4 weeks as one cycle) and adalimumab (administered once every 4 weeks, with 4 weeks as one cycle). After completing 2 cycles of treatment, they were sequentially given liposomal irinotecan combined with 5-FU/LV, oxaliplatin (administered once every 2 weeks, with 4 weeks as one cycle) and adalimumab (administered once every 4 weeks, with 4 weeks as one cycle). After completing 2 cycles of sequential treatment, surgical evaluation was conducted: for patients who could undergo radical surgical resection, surgery was performed within 2-4 weeks after the end of the conversion treatment stage, and the postoperative treatment plan was selected based on the investigator's judgment; for patients who could not undergo radical surgical resection, subsequent treatment plans could be selected based on the investigator's judgment.

SUMMARY:
The goal of this interventional study is to learn about the clinical efficacy of sequential therapy (albumin paclitaxel, gemcitabine combined with PD-L1 antibodies, followed by liposomal irinotecan, oxaliplatin and 5-FU/LV combined with PD-L1 antibodies). The main questions it aims to answer are:

Does the sequential therapy increase the resection rate of borderline resectable / locally advanced pancreatic cancer? Does the sequential therapy represent an effective and safe treatment? Participants will receive two distinct chemotherapy regimens, each combined with a PD-L1 antibody, administered in sequence for two cycles each.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old, gender not restricted
* According to the NCCN Clinical Practice Guidelines for Pancreatic Cancer (2024.V2 version), patients with borderline resectable/locally advanced pancreatic cancer as evaluated by multidisciplinary and imaging assessment, the definition of borderline resectability includes:

  1. No distant metastasis;
  2. Arteries: 1. Pancreatic head/neck: The tumor is in contact with the common hepatic artery and does not extend to the abdominal aorta or the hepatic artery bifurcation, and can be safely resected and reconstructed; the tumor is in contact with the superior mesenteric artery ≤ 180°; the tumor contacts variant arteries (such as the accessory right hepatic artery, replacement of the hepatic right artery, replacement of the common hepatic artery or the starting part of the accessory/secondary artery, etc.), but can be safely resected and reconstructed. 2. Pancreatic body/tail: The tumor is in contact with the abdominal aorta ≤ 180°;
  3. Veins: The tumor is in contact with the superior mesenteric vein or portal vein > 180°, or contact ≤ 180° combined with irregular venous contour or venous thrombosis, and there are appropriate blood vessels at the proximal and distal ends of the affected area that can be completely resected and reconstructed; the tumor contacts the inferior vena cava;

     Local advanced pancreatic cancer is defined as:

  <!-- -->

  1. No distant metastasis;
  2. Arteries: 1. Pancreatic head/neck: The tumor is in contact with the superior mesenteric artery or the celiac trunk artery > 180°; 2. Pancreatic body/tail: The tumor is in contact with the superior mesenteric artery or the celiac trunk artery > 180°; the tumor contacts the celiac trunk artery and invades the abdominal aorta;
  3. Veins: Due to tumor invasion, vein occlusion or involvement of a large area of the superior mesenteric vein and ileal branch, it is impossible to safely reconstruct the portal vein - superior mesenteric vein;
* No previous anti-tumor treatment (including radiotherapy, ablation, chemotherapy, targeted therapy, immunotherapy, etc.), investigational drug treatment;
* Must have at least one measurable lesion as the target lesion (according to RECIST v1.1 standard);
* ECOG: 0 - 1
* Expected survival ≥ 3 months;
* Good function of major organs, that is, in accordance with the following standards (within 14 days before randomization, no blood components, cell growth factors were received):

  1. Neutrophils ≥ 1.5 * 10^9/L; platelets ≥ 80 * 10^9/L; hemoglobin ≥ 9 g/dl; serum albumin ≥ 3 g/dl;
  2. Total bilirubin ≤ 1.5 times the upper limit of normal (biliary obstruction allows biliary drainage); ALT and AST ≤ 3 times the upper limit of normal;
  3. Serum creatinine ≤ 1.5 times the upper limit of normal, creatinine clearance rate ≥ 60 ml/min;
  4. INR ≤ 1.5 times the upper limit of normal and APTT ≤ 1.5 times the upper limit of normal (for those using stable doses of anticoagulation therapy such as low molecular weight heparin or warfarin and INR within the expected treatment range of the anticoagulant can be screened);
  5. Electrocardiogram: QTcF ≤ 450 ms (male), ≤ 470 ms (female);
  6. Cardiac echocardiography: LVEF (left ventricular ejection fraction) ≥ 50%;
* Female participants with reproductive capacity must undergo a blood pregnancy test 3 days before the first administration, and the result must be negative, not in lactation period, and willing to take effective contraceptive methods during the trial and within 2 months after the last administration of ademetelstat or 9 months after chemotherapy drugs (whichever is longer) (for male participants whose partners have reproductive capacity, surgical sterilization should be performed, or agree to take effective contraceptive methods within 2 months after the last administration of ademetelstat or 6 months after chemotherapy drugs, during the study period, sperm donation is not allowed).
* Participants voluntarily join this study and sign the informed consent form.

Exclusion Criteria:

* Pancreatic cancer originating from non-pancreatic ductal epithelium, including pancreatic neuroendocrine carcinoma, pancreatic acinar cell carcinoma, pancreatic blastoma, solid-pseudopapillary tumors patients
* Patients with known central nervous system metastasis
* Severe gastrointestinal dysfunction (with bleeding, obstruction; grade 2 or higher inflammation; grade 1 or higher diarrhea)
* Randomly within the previous 2 weeks, there was third-space effusion (such as large pleural effusion) that could not reach a stable state (after removing the drainage tube, no intervention treatment was required)
* Abdominal effusion with clinical symptoms, requiring puncture and drainage, or patients who had undergone abdominal effusion drainage within 3 months previously (excluding those with only imaging showing a small amount of abdominal effusion and controllable, but without clinical symptoms)
* Currently accompanied by interstitial pneumonia or interstitial lung disease, or having a history of interstitial pneumonia or interstitial lung disease requiring hormone treatment previously, or other possible pulmonary fibrosis, organizing pneumonia (such as obliterative bronchiolitis), pneumoconiosis, drug-related pneumonia, idiopathic pneumonia or in the screening period, chest CT showing active pneumonia or severely impaired lung function subjects; active tuberculosis
* Presence of active autoimmune disease or having a history of autoimmune disease that may recur [including but not limited to autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, pituitary inflammation, vasculitis, nephritis, hyperthyroidism, hypothyroidism (only subjects with controlled hormone replacement therapy can be enrolled)], having a skin disease that does not require systemic treatment such as vitiligo, psoriasis, alopecia, receiving insulin treatment for controlled type 1 diabetes or having completely resolved childhood asthma and no need for any intervention after adulthood, eligible for enrollment
* Known peripheral neuropathy (CTCAE ≥ 3 grade)
* Known dihydroorotate dehydrogenase (low activity) or deficiency
* Randomly within the previous 2 weeks, had severe infection (CTCAE > 2 grade), such as severe pneumonia requiring hospitalization, sepsis, infection complications, etc.; randomly within the previous 2 weeks, had symptoms and signs of infection requiring intravenous antibiotic treatment (except for prophylactic use of antibiotics)
* Had received any of the following treatments:

  1. Randomly within the previous 2 weeks, the medication used included strong inhibitors/inducers of CYP3A4, CYP2C8 or strong inhibitors of UGT1A1;
  2. Randomly within the previous 2 weeks, received immunosuppressants or systemic hormone treatment to achieve immunosuppression purposes (dose > 10mg/day prednisone or other equivalent efficacy hormones);
  3. Randomly within the previous 2 weeks, received radiotherapy;
  4. Randomly within the previous 4 weeks, underwent major surgery (such as thoracotomy, laparotomy, etc.);
  5. Randomly within the previous 4 weeks, received any other clinical research drug treatment, unless it is an observational (non-interventional) clinical study or follow-up of an interventional clinical study.
* Abnormal coagulation function, with bleeding tendency or undergoing thrombolysis or anticoagulation treatment. Allowed to use preventive low-dose aspirin (≤100mg/day) or low-molecular-weight heparin (enoxaparin 40mg/day and other low-molecular-weight heparins at equivalent doses)
* Had poor control of clinical symptoms or diseases of the heart, such as: (1) NYHA grade 2 or above heart failure; (2) unstable angina pectoris; (3) having had a myocardial infarction within 6 months; (4) having clinical significance of supraventricular or ventricular arrhythmias and requiring treatment or intervention
* Randomly within the previous 5 years had malignant tumors other than pancreatic cancer, except for adequately treated cervical carcinoma in situ, basal cell or squamous cell carcinoma of the skin
* Those who are known to be allergic to PD-L1, gemcitabine, albumin paclitaxel, gemcitabine, albumin paclitaxel, irinotecan liposome, other liposome products, oxaliplatin, 5-FU, folic acid calcium, or any of the components in the above products
* Those who are known to have acquired immunodeficiency syndrome (AIDS) or have tested positive for HIV, or active syphilis patients
* Those who have a clear history of neurological or mental disorders, including epilepsy or dementia
* Based on the investigator's judgment, the subjects have other factors that may cause them to be forced to terminate the study prematurely, such as non-compliance with the protocol, having other serious diseases (including mental disorders) that require combined treatment, having severely abnormal laboratory test values with clinical significance, family or social factors, and situations that may affect the safety of the subjects or the collection of trial data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Estimated)
Dates: Start 2025-10-10 (Estimated); Primary Completion 2026-04-09 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
18-month overall survival (OS) rate | From the date of first enrollment to 18 months later.
  To test whether the 18-month OS rate of patients with borderline resectable or locally advanced pancreatic cancer treated with the sequential therapy was comparable to that of the historical data of the general adult population.

SECONDARY OUTCOMES:
Surgical conversion rate | From the date of first enrollment to the date of completion of follow-up of the last patient, up to 30 months.
  The surgical conversion rate refers to the process of transforming an initially inoperable tumor into one that can be removed through a pre-defined treatment plan. The conversion rate is the proportion of subjects who successfully underwent the conversion treatment among all subjects who received such treatment.
Overall survival rate (OS) | From the date of first enrollment to the date of completion of follow-up of the last patient, up to 30 months.
Event-free survival (EFS) | From the date of first enrollment to the date of completion of follow-up of the last patient, up to 30 months.
  Survival time from the first enrollment to the date of first documented progression or the date of death.
R0 resection rate | From the date of first enrollment to the date of completion of follow-up of the last patient, up to 30 months.
  The R0 resection rate is defined as the proportion of subjects who were assessed as having achieved R0 resection (complete tumor removal, with no cancer cells found at the microscopic margin, no cancer cells remaining either macroscopically or under the microscope, and the lesion was completely removed) after the surgery.
R1 resection rate | From the date of first enrollment to the date of completion of follow-up of the last patient, up to 30 months.
  The R1 resection rate is defined as the proportion of subjects who were assessed as having undergone R1 resection (microscopic residual, all large lesions were removed, and there were cancer cells at the microscopic margin) after the surgery.
Objective response rate (ORR) | From the date of first enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 30 months.
  ORR is defined as the percentage of patients who achieve complete response (CR) or partial response (PR) based on the Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1.
Toxicity and side effects and tolerability assessment | From the date of first therapy administration to within 90 days, up to 30 months.
  Safety and tolerance will be evaluated by incidence, severity and outcomes of adverse events (AEs) and categorized by severity in accordance with the NCI CTCAE Version 5.0.

IPD SHARING:
Plan to Share IPD: No